CLINICAL TRIAL: NCT05298683
Title: A Phase 2 Study of Isatuximab in Combination With Pomalidomide and Dexamethasone in MM Patients Who Received One Prior Line of Therapy Containing Lenalidomide and a Proteasome Inhibitor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAE115
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma; Renal Impairment; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases | interventions — isatuximab; pomalidomide; Dexamethasone; Acetaminophen; Ranitidine; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): Eligible patients will initially receive six 28-day cycles of isatuximab, pomalidomide, and low-dose dexamethasone. Patients will be allowed to continue treatment until disease progression, death, unacceptable AEs, lost to follow-up, or consent withdrawal.
  Isatuximab will be given at a dose of 10 mg/kg QW by IV infusion.
  Pomalidomide will be given at 4 mg orally(PO) on Days 1-21 of each cycle.
  Dexamethasone will be given at 40 mg (20 mg for ≥75 years old) PO, or IV on days 1, 8, 15, and 22 in each cycle.
  Acetaminophen (paracetamol) will be given at 650-1000 mg PO 15-30 minutes (but no longer than 60 minutes) before isatuximab infusion.
  Ranitidine or equivalent will be given at 50 mg 15-30 minutes (but no longer than 60 minutes) before isatuximab infusion.
  Diphenhydramine or equivalent will be given at 25-50 mg 15-30 minutes (but no longer than 60 minutes) before isatuximab infusion.
  Interventions: Drug: Isatuximab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Acetaminophen (paracetamol); Drug: Ranitidine (or equivalent); Drug: Diphenhydramine (or equivalent)

INTERVENTIONS:
Drug: Isatuximab — Intravenous (IV) infusion. Dose regimen: Isatuximab will be given at a dose of 10 mg/kg QW by IV infusion on Days 1, 8, 15, and 22 in Cycle 1 and Days 1 and 15 in subsequent cycles. In patients with ≥VGPR who will be randomized to receive isatuximab once monthly from Cycle 7, isatuximab will be given on day 1 of each cycle.
Drug: Pomalidomide — Route of administration: Oral (PO). Dose regimen: Pomalidomide will be given at 4 mg orally (PO) will be given on Days 1-21 of each cycle.
Drug: Dexamethasone — Route of administration: PO or IV. Dose regimen: Dexamethasone will be given at 40 mg (20 mg for ≥75 years old) PO, or IV will be given on days 1, 8, 15, and 22 in each cycle.
Drug: Acetaminophen (paracetamol) — Route of administration: PO. Dose regimen: Acetaminophen (paracetamol) will be given at 650-1000 mg PO 15-30 minutes (but no longer than 60 minutes) before isatuximab infusion
Drug: Ranitidine (or equivalent) — Route of administration: IV. Dose regimen: Ranitidine or equivalent will be given at 50 mg 15-30 minutes (but no longer than 60 minutes) before isatuximab infusion.
Drug: Diphenhydramine (or equivalent) — Route of administration: IV. Dose regimen: Diphenhydramine or equivalent will be given at 25-50 mg 15-30 minutes (but no longer than 60 minutes) before isatuximab infusion.

SUMMARY:
This is an investigator-initiated (IIS), phase 2, prospective, open-label, multinational study, designed to be conducted in approximately 14 sites. Eligible patients will initially receive six 28-day cycles of isatuximab, pomalidomide, and low-dose dexamethasone.

Following this phase:

Patients who achieve ≥VGPR will be randomized in a 1:1 ratio to receive isatuximab, given either Q2W or once monthly, plus pomalidomide and low-dose dexamethasone.

Patients with <VGPR will continue treatment with isatuximab Q2W, pomalidomide, and low-dose dexamethasone.

The study will last for 42 months (recruitment and follow-up period), starting from the date of the first patient in (FPI) to the date of the last patient last visit (LPLV).

Core study procedures consist of baseline and post-baseline safety and disease evaluations, including physical examination, hematologic/clinical chemistry tests, radiologic assessments, bone marrow evaluations, and blood/urine M-protein assessments.

Patients will be allowed to continue treatment until disease progression, death, unacceptable AEs, lost to follow-up, or consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed an informed consent form (ICF) indicating that he or she understands the purpose of the procedures required for the study and are willing to participate in the study. Patients must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.
2. Male or female patients aged 18 years or older at the time of the ICF signature.
3. Patients who have received ONLY one prior line of anti-myeloma therapy, which included lenalidomide (at least 2 cycles, either alone or in combination) and a proteasome inhibitor (e.g. bortezomib, carfilzomib, ixazomib). Patients must have achieved at least a response of MR or better based on the investigator's determination of response as defined by the IMWG criteria.

   Note:

   An induction treatment followed by ASCT and consolidation/maintenance will be considered as one line of treatment.
4. Patients with a documented diagnosis of MM and with current evidence of measurable disease defined as:

   * Serum monoclonal protein (M-protein) level ≥0.5 g/dL, measured using serum protein electrophoresis (SPEP) and/or
   * Urine M-protein level ≥200 mg/24 hours, measured using urine protein electrophoresis (UPEP), or
   * Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
5. Patients must have documented evidence of PD, based on the investigator's determination of response as defined by the IMWG criteria, on or after the last line of treatment.
6. Adequate bone marrow and hepatic function as defined by ALL the laboratory criteria:

   * Absolute Neutrophil Count (ANC) ≥1.0 x 109/L; GCSF administration is not allowed to reach this level
   * Hemoglobin level ≥7.5 g/dL (≥4.65 mmol/L);
   * Platelet count ≥75 x 109/L in patients in whom <50% of bone marrow nucleated cells are plasma cells OR Platelet count ≥50 x 109/L in patients in whom ≥50% of bone marrow nucleated cells are plasma cells; [transfusions are not permitted to reach this level]
   * Alanine aminotransferase (ALT) level ≤2.5 x ULN
   * Aspartate aminotransferase (AST) level ≤2.5 x ULN
   * Total bilirubin level ≤1.5 x ULN (except for Gilbert Syndrome: direct bilirubin ≤1.5 x ULN)
   * Creatinine clearance ≥30 mL/min; calculated using Cockcroft Gault
   * Serum calcium corrected for albumin ≤14.0 mg/dL (≤3.5 mmol/L), or free ionized calcium ≤ 6.5 mg/dL (≤1.6 mmol/L)
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2
8. For patients experiencing toxicities resulting from previous therapy, the toxicities must be resolved or stabilized to ≤ Grade 1.

Exclusion Criteria:

1. Previous therapy with any anti-CD38 monoclonal antibody.
2. Previous exposure to pomalidomide.
3. Patient has received anti-myeloma treatment within two weeks or five pharmacokinetic half-lives of the treatment, whichever is longer, before Cycle 1, Day 1 (C1D1). The only exception is emergency use of a short course of corticosteroids (the equivalent of dexamethasone 40 mg/day for a maximum of 4 days) for palliative treatment before C1D1.
4. Previous allogeneic stem cell transplant or autologous stem cell transplantation (ASCT) within 12 weeks before C1D1.
5. History of malignancy (other than MM) within three years before C1D1 (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesions that in the opinion of the investigator, with concurrence with the Sponsor's medical monitor, is considered cured with minimal risk of recurrence within three years).
6. Clinical signs of meningeal involvement of MM.
7. Clinically significant cardiac disease, including:

   1. Myocardial infarction within six months before C1D1, or unstable or uncontrolled condition (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
   2. Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Grade 3 or higher) or clinically significant electrocardiogram (ECG) abnormalities.
   3. Electrocardiogram showing a baseline QT interval as corrected QTc >470 msec.
8. Known:

   1. Active hepatitis A
   2. To be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Patients with resolved infection (i.e., patients who are positive for antibodies to hepatitis B core antigen [antiHBc] and/or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Patients with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
   3. To be seropositive for hepatitis C (defined by a positive test for Hepatitis C virus (HCV) antibodies. A positive HCV antibody test should be confirmed by a HCV RNA test. EXCEPTION: Patients in the setting of a sustained virologic response, defined as aviremia at least 12 weeks after completion of antiviral therapy, are not excluded).
9. Known to be seropositive for human immunodeficiency virus (defined by positive testing for human immunodeficiency virus (HIV) antibodies).
10. Gastrointestinal disease that may significantly alter the absorption of pomalidomide.
11. Patient has plasma cell leukemia (>2.0 × 109/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
12. Any concurrent medical or psychiatric condition or disease (e.g., active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results or that, in the opinion of the investigator, would constitute a hazard for participating in this study.
13. Ongoing ≥Grade 2 peripheral neuropathy.
14. Patient had ≥Grade 3 rash during prior therapy.
15. Patient has had major surgery within two weeks before C1D1, or has not fully recovered from an earlier surgery, or has a surgery planned during the time the patient is expected to participate in the study or within two weeks after the last dose of study drug administration. Note: patients with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery.
16. Patient has known allergies, hypersensitivity, or intolerance to any of the study drugs, monoclonal antibodies, human proteins, or their excipients (refer to isatuximab IB) or known sensitivity to mammalian-derived products.
17. Patient was vaccinated with live vaccines within four weeks prior to C1D1.
18. Pregnant or nursing women.
19. a. Females of childbearing potential (FCBP) unwilling to prevent pregnancy with the use of two reliable methods of contraception for ≥4 weeks before the start of study treatment, during treatment (including dose interruptions), and up to five months following the last dose of isatuximab or three months following the last dose of the rest of the study treatment, whichever is longer. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap).

    b. FCBP who are unwilling or unable to be tested for pregnancy: a) before study treatment initiation, b) weekly during 1st month of treatment and then prior to each treatment cycle administration or c) every two weeks in case of irregular menstrual cycles, and d) up to five months following the last dose of isatuximab or three months following the last dose of the rest of the study treatment, whichever is longer.
20. Male participants who refuse to practice true abstinence or use a condom during sexual contact with a pregnant female or an FCBP while participating in the study, during dose interruptions and at least five months following the last dose of isatuximab or three months following the last dose of the rest of the study treatment, whichever is longer, even if he has undergone a successful vasectomy.

Note 1: an FCBP is a female who: 1) has achieved menarche at some time point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Note 2: True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | After six months of treatment with isatuximab plus pomalidomide and low-dose dexamethasone
  The primary endpoint is the ORR after six months of treatment with isatuximab in combination with pomalidomide, and low-dose dexamethasone. ORR is defined as the proportion of patients with stringent complete response (sCR), complete response (CR), VGPR, and partial response (PR), as assessed by the Investigator using the IMWG response criteria.

SECONDARY OUTCOMES:
Progression-free Survival | From study treatment initiation to progressive disease (PD), or initiation of further anti-myeloma treatment, or death, whichever occurs first. Maximum time period 42 months.
  Defined as the time from study treatment initiation (Cycle 1 Day 1) to the date of first documentation of progressive disease (PD), as assessed by the Investigator using the IMWG response criteria, or the date of death from any cause, or the initiation of further anti-myeloma treatment, or data cut-off, whichever occurs first.
Overall Survival (OS) | From study treatment initiation to death. Maximum time period 42 months.
  Defined as the time from study treatment initiation (Cycle 1 Day 1) to the date of death from any cause. OS will be assessed throughout the treatment period and post EOT during long term follow-up until the end of the study.
Minimal Residual Response (MRD) | Through study completion. Maximum time 42 months.
  Defined as the proportion of patients achieving MRD-negative status, assessed at CR.
Time to Response (TTR) | From study treatment initiation to partial response (PR), or better. Maximum time period 42 months.
  Defined as the time from study treatment initiation (Cycle 1, Day 1) to the date of the first objective response of PR or better.
Duration of Response (DoR) | From time response is achieved to progressive disease (PD), or death, whichever comes first. Maximum time period 42 months.
  Defined as the time from the date of the first response, as determined by the Investigator, to the date of the first PD (based on the International Myeloma Working Group [IMWG] response criteria) or death, whichever occurs first. DoR will be determined only for patients who have achieved ≥PR.
Safety | Study treatment initiation until 30 days after last study treatment. Maximum time period 42 months.
  i.e. Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof, Principal Investigator — Department of Clinical Therapeutics, School of Medicine, National Kapodistrian University of Athens (NKUA)
Locations (6):
- Greece (6):
  - General Hospital of Athens "Evangelismos", Athens
  - Anticancer Oncology Hospital of Athens "Agios Savvas", Athens
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patra, Pátrai
  - Anticancer Hospital of Thessaloniki "Theageneio", Thessaloniki